CLINICAL TRIAL: NCT00172614
Title: The Roles of Cytokines in the Mechanism of Insulin Resistance and Energy Balance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701201
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-29 (Estimated); Status verified 2004-12

CONDITIONS: Metabolic Syndrome X; Cachexia; Insulin Resistance
Keywords: metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Cachexia; Insulin Resistance

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Insulin resistance and disturbances in energy homeostasis are associated with body weight changes, such as diabetes, hypertension, hyperlipidemia, obesity, cancer cachexia, aging, and acute or chronic infectious diseases. Cytokines secreted by adipose tissue and inflammatory cells play important roles in the pathological conditions. Several novel cytokines were disclosed recently, but their functions have not been well known. Further investigation of these cytokines, resulting in insulin resistance and energy homeostasis, is very important to elucidate the mechanisms and develop new therapeutic strategies.

DETAILED DESCRIPTION:
We are studying patients with body weight change, increased or decreased. Healthy people are the control group. We are recording body weight, body height, and physical exam results. In addition, we are drawing peripheral blood for further biochemical and cytokine assays.

ELIGIBILITY:
Inclusion Criteria:

* Insulin resistance condition

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Shiun Tsai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan